CLINICAL TRIAL: NCT03643835
Title: Efficacy of an Investigational Thermal Rehab Machine on Body Cooling in Hyperthermic Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Greensboro (Other)
Collaborators: Statim Technologies, LLC (Unknown)
Responsible Party: Principal Investigator, William Adams, Assistant Professor, University of North Carolina, Greensboro
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Device Feasibility
Other Study IDs: 18-0280
Record Dates: First submitted 2018-08-15; First posted 2018-08-23 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Cryotherapy Effect

STUDY DESIGN:
Intervention Model Description: Participants will complete three trials under three different body cooling conditions/interventions; passive cooling using the body's natural body cooling mechanisms, body cooling using forearm ice towels, and cooling using the investigational thermal rehab machine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Thermal rehab machine (Experimental): Participants, following exercise-induced hyperthermia, will be cooled using a Thermal Rehab Machine (Polar Breeze, Statim Technologies, LLC, Clearwater Florida), which is a micro-environmental air chiller. The device will be placed over the subjects head and through trans pulmonary cooling, will cool the body.
  Interventions: Device: Thermal Rehab Machine
- Forearm Ice Towels (Active Comparator): Participants, following exercise-induced hyperthermia, will be cooled using forearm ice towels. Cotton-blend towels will be doused in ice-water and then wrapped around participant's forearms (elbow to wrist). The towels will be rotated (re-wetted) every 2 minutes)
  Interventions: Other: Forearm Ice Towels
- Passive Cooling (No Intervention): Participants, following exercise-induced hyperthermia, will undergo a period of passive rest to allow the body to cool via natural mechanisms of evaporation of sweat from the skin's surface and convection

INTERVENTIONS:
Device: Thermal Rehab Machine — The Polar Breeze unit is a microenvironmental air-chiller. That means it is a single-pass air-conditioner capable of cooling external air
  Other Names: Polar Breeze
  Arms: Thermal rehab machine
Other: Forearm Ice Towels — Towels that are wetted with ice water and wrapped around participants forearms (length of arm from wrist to elbow)
  Arms: Forearm Ice Towels

SUMMARY:
Exertional heat stroke (EHS) is an emergency medical condition that is prevalent in military soldiers, athletes, and laborers. It is diagnosed when the rectal temperature is above 40°C with the presence of central nervous dysfunction (altered mental status). The gold standard method of care for EHS is immediate onsite whole body cooling using cold-water immersion (cooling rates >0.15°C•min-1), which is reported to have the highest cooling rate. In the treatment of EHS, selecting a cooling modality with a high cooling rate becomes crucial to minimize the time above the critical threshold of body temperature at 40°C to less than 30 minutes for the best chance of survival and to minimize the severity of prognosis. However, in situations where cold water immersion is not feasible (in certain military, firefighter, or other remote settings), other cooling modalities must be available that have a cooling capacity similar to that of cold-water immersion. In this proposed study, the investigators aim to examine the cooling rates of the Polar Breeze® device (developed by Statim Technologies, LLC, Clearwater, FL) compared to rotating ice towels, a cooling method often recommended by sports medicine professionals as an alternative to cold-water immersion, and passive rest in participants with exercise-induced hyperthermia.

ELIGIBILITY:
Inclusion Criteria:

* male between the ages of 18-35.
* recreationally active (regularly exercise at a minimum of 4-5 times per week for greater than 30 minutes per session)

Exclusion Criteria:

* chronic health problems,
* fever or current illness at the time of testing
* history of cardiovascular, metabolic, or respiratory disease
* current musculoskeletal injury that limits physical activity
* history of exertional heat illness in the past three years.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Internal Body Temperature | 0, 5, 10, 15, 20, 25, 30, 35, 40, 45, 50, 55, 60 minutes post onset of cooling
  The rate at which body temperature is reduced during whole body cooling following exercise-induced hyperthermia.

CONTACTS AND LOCATIONS:
Overall Officials: William M Adams, PhD, Principal Investigator — University of North Carolina, Greensboro
Locations (1):
- University of North Carolina at Greensboro, Greensboro, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2018-08-15): https://cdn.clinicaltrials.gov/large-docs/35/NCT03643835/ICF_000.pdf